CLINICAL TRIAL: NCT02769338
Title: Protocol-guided Rapid Evaluation of Veterans Experiencing New Transient Neurological Symptoms (PREVENT) (QUE 15-280)
Brief Title: Protocol-guided Rapid Evaluation of Veterans Experiencing New Transient Neurological Symptoms
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 16-006
Record Dates: First submitted 2016-04-28; First posted 2016-05-11 (Estimated); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-03

CONDITIONS: Transient Ischemic Attack; Stroke
Keywords: Implementation; Quality Improvement; Stroke; Transient Ischemic Attack; TIA; Systems Redesign; QI Intervention
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke

STUDY DESIGN:
Intervention Model Description: Stepped-wedge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QI with External Facilitation (Experimental): Receive external facilitation to support implementation of the quality improvement program
  Interventions: Other: Quality Improvement Program
- Control (No Intervention): Non-Intervention VA Medical Centers

INTERVENTIONS:
Other: Quality Improvement Program — The Intervention is a QI Program that will include multiple components as described above.
  Other Names: QI Intervention
  Arms: QI with External Facilitation

SUMMARY:
This program will seek to implement a quality improvement program to improve the care of Veterans with TIA or minor stroke at 6 Veteran Health Administration Hospitals. The investigators will evaluate the implementation and effectiveness of the quality improvement program.

DETAILED DESCRIPTION:
Aim 1. To develop a quality improvement program to improve the care of Veterans with TIA or minor stroke that can be deployed nationwide. The program will include multiple components: a reporting system that is based on validated electronic quality measures (eCQMs) that will allow staff to monitor the time-sensitive processes of care and outcomes of their population of Veterans with TIA or minor stroke; clinical protocols to improve the timeliness and completeness of care; professional education materials; and clinical note templates for use by nursing and pharmacy staff. Lessons learned at the individual sites engaged in the quality improvement program will be shared across sites by use of a web-based platform and a virtual collaborative. We will assess end user's assessment of the program and its core elements.

Aim 2. To evaluate the effectiveness of the Aim 1 QI intervention program for Veterans with TIA or minor stroke against usual care. Teams at the 6 intervention sites will be given the quality improvement program components. The primary effectiveness outcome is the proportion of Veterans who received all of the guideline-concordant processes of care for which they are eligible referred to as the "Without-Fail" care rate.

Aim 3. To evaluate the implementation of the QI intervention program across the 6 participating sites. The two primary implementation outcomes will be the number of implementation activities completed during the one-year active implementation period and the final level of team organization (defined as the Group Organization (GO Score)) for improving TIA care at the end of the 12-month active implementation period.

Secondary Aim To evaluate the sustainability of the program. Sustainability will be evaluated over a one-year period that begins immediately after the one-year active implementation period. We will compare the Without-Fail rate in the sustainability period to the baseline period and the post-implementation period.

ELIGIBILITY:
Inclusion Criteria:

* This program will seek VA hospitals that are self-designated as either a VHA Primary Stroke Center or a Limited Hours Stroke Facility or Supporting Stroke Center.
* Eligibility for staff interviews is based on involvement in the QI intervention and willingness to participate.

Exclusion Criteria:

* Unwilling to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2292 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M. Bravata, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN; Teresa M. Damush, PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Investigators interested in examining PREVENT project data should contact the PI, Dr. Dawn Bravata.

REFERENCES:
- [Background] Penney LS, Homoya BJ, Damush TM, Rattray NA, Miech EJ, Myers LJ, Baird S, Cheatham A, Bravata DM. Seeding Structures for a Community of Practice Focused on Transient Ischemic Attack (TIA): Implementing Across Disciplines and Waves. J Gen Intern Med. 2021 Feb;36(2):313-321. doi: 10.1007/s11606-020-06135-z. Epub 2020 Sep 1. PMID 32875499
- [Background] Rattray NA, Damush TM, Miech EJ, Homoya B, Myers LJ, Penney LS, Ferguson J, Giacherio B, Kumar M, Bravata DM. Empowering Implementation Teams with a Learning Health System Approach: Leveraging Data to Improve Quality of Care for Transient Ischemic Attack. J Gen Intern Med. 2020 Nov;35(Suppl 2):823-831. doi: 10.1007/s11606-020-06160-y. Epub 2020 Sep 1. PMID 32875510
- [Background] Li J, Zhang Y, Myers LJ, Bravata DM. Power calculation in stepped-wedge cluster randomized trial with reduced intervention sustainability effect. J Biopharm Stat. 2019;29(4):663-674. doi: 10.1080/10543406.2019.1633658. Epub 2019 Jul 18. PMID 31317805
- [Background] Bravata DM, Myers LJ, Homoya B, Miech EJ, Rattray NA, Perkins AJ, Zhang Y, Ferguson J, Myers J, Cheatham AJ, Murphy L, Giacherio B, Kumar M, Cheng E, Levine DA, Sico JJ, Ward MJ, Damush TM. The protocol-guided rapid evaluation of veterans experiencing new transient neurological symptoms (PREVENT) quality improvement program: rationale and methods. BMC Neurol. 2019 Nov 20;19(1):294. doi: 10.1186/s12883-019-1517-x. PMID 31747879
- [Result] Bravata DM, Myers LJ, Perkins AJ, Zhang Y, Miech EJ, Rattray NA, Penney LS, Levine D, Sico JJ, Cheng EM, Damush TM. Assessment of the Protocol-Guided Rapid Evaluation of Veterans Experiencing New Transient Neurological Symptoms (PREVENT) Program for Improving Quality of Care for Transient Ischemic Attack: A Nonrandomized Cluster Trial. JAMA Netw Open. 2020 Sep 1;3(9):e2015920. doi: 10.1001/jamanetworkopen.2020.15920. PMID 32897372
- [Result] Damush TM, Miech EJ, Rattray NA, Homoya B, Penney LS, Cheatham A, Baird S, Myers J, Austin C, Myers LJ, Perkins AJ, Zhang Y, Giacherio B, Kumar M, Murphy LD, Sico JJ, Bravata DM. Implementation Evaluation of a Complex Intervention to Improve Timeliness of Care for Veterans with Transient Ischemic Attack. J Gen Intern Med. 2021 Feb;36(2):322-332. doi: 10.1007/s11606-020-06100-w. Epub 2020 Nov 3. PMID 33145694
- [Result] Damush TM, Penney LS, Miech EJ, Rattray NA, Baird SA, Cheatham AJ, Austin C, Sexson A, Myers LJ, Bravata DM. Acceptability of a complex team-based quality improvement intervention for transient ischemic attack: a mixed-methods study. BMC Health Serv Res. 2021 May 12;21(1):453. doi: 10.1186/s12913-021-06318-2. PMID 33980224
- [Derived] Baird SA, Damush TM, Rattray NA, Penney LS, Miech EJ, Homoya BJ, Ferguson J, Myers LJ, Bravata DM. Using a "Kickoff" to build implementation partner teams and action plans for active implementation of a quality improvement project. Front Health Serv. 2025 Jun 10;5:1580653. doi: 10.3389/frhs.2025.1580653. eCollection 2025. PMID 40556841
- [Derived] Myers LJ, Perkins AJ, Zhang Y, Bravata DM. Identifying transient ischemic attack (TIA) patients at high-risk of adverse outcomes: development and validation of an approach using electronic health record data. BMC Neurol. 2022 Jul 12;22(1):256. doi: 10.1186/s12883-022-02776-1. PMID 35820867
- [Derived] Bravata DM, Miech EJ, Myers LJ, Perkins AJ, Zhang Y, Rattray NA, Baird SA, Penney LS, Austin C, Damush TM. The Perils of a "My Work Here is Done" perspective: a mixed methods evaluation of sustainment of an evidence-based intervention for transient ischemic attack. BMC Health Serv Res. 2022 Jul 4;22(1):857. doi: 10.1186/s12913-022-08207-8. PMID 35787273
- [Derived] Penney LS, Damush TM, Rattray NA, Miech EJ, Baird SA, Homoya BJ, Myers LJ, Bravata DM. Multi-tiered external facilitation: the role of feedback loops and tailored interventions in supporting change in a stepped-wedge implementation trial. Implement Sci Commun. 2021 Jul 27;2(1):82. doi: 10.1186/s43058-021-00180-3. PMID 34315540

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: VA hospitals
Period: Baseline Period
Arm/Group | QI With External Facilitation | Control
Started | 162; 6 VA hospitals | 973; 36 VA hospitals
Completed | 162; 6 VA hospitals | 973; 36 VA hospitals
Not Completed | 0; 0 VA hospitals | 0; 0 VA hospitals
Period: Active Implementation Period
Arm/Group | QI With External Facilitation | Control
Started | 189; 6 VA hospitals (As described in the baseline characteristics tab, there were 6 PREVENT intervention sites and 36 control sites. Different patients were cared for at these sites during the baseline period versus the active implementation period: PREVENT Intervention baseline N=162, intervention implementation N=189; control baseline N=973, control implementation N=968.) | 968; 36 VA hospitals
Completed | 189; 6 VA hospitals | 968; 36 VA hospitals
Not Completed | 0; 0 VA hospitals | 0; 0 VA hospitals

BASELINE CHARACTERISTICS:
Population: There were 6 intervention sites and 36 control sites and two time periods (baseline and active implementation). Different patients were cared for at the sites during the two time periods. During baseline, there were N=162 PREVENT intervention patients and N=973 patients at control sites. During the active implementation period, there were N=189 patients at PREVENT intervention sites and N=968 at control sites.
Units Other Than Participants: Number of units (VA hospitals)
Groups:
- Total: Total of all reporting groups
Arm/Group | QI With External Facilitation | Control | Total
Number analyzed (Participants) | 162 | 973 | 1135
Number analyzed (Number of units (VA hospitals)) | 6 | 36 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (11.2) | 71.7 (11.3) | 71.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 53 | 61
  Male | 154 | 920 | 1074
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 45 | 63
  Not Hispanic or Latino | 144 | 928 | 1072
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 145 | 182
  White | 116 | 770 | 886
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 49 | 57
The Without-Fail Rate [Count of Participants; unit: Participants] — Population: Not all patients were eligible for the process measures that were included in the without-fail rate.
  Participants
    number analyzed (Participants) | 158 | 893 | 1051
    (all) | 58 | 345 | 403

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness: Without-fail Care Rate
Description: Teams at the 6 intervention sites will be given both the QI program (to improve care) and eCQM data (to monitor the care they are delivering to their patients). The primary effectiveness outcome is the proportion of Veterans who received all of the guideline-concordant processes of care for which they are eligible referred to as the "Without-Fail" care rate. Determined by analysis of electronic medical record data.
Time Frame: Over the course of One Year active implementation
Population: During the active implementation period, there were N=189 patients at the intervention sites, 176 of whom were eligible for the without-fail measure; and there were N=968 patients at the control sites, 869 of whom were eligible for the without-fail measure.
Measure: Count of Participants; unit: Participants
Arm/Group | QI With External Facilitation | Control
Number analyzed (Participants) | 176 | 869
Participants | 95 | 363

2. Secondary Outcome: Recurrent Vascular Events
Description: The recurrent event endpoint included: congestive heart failure, myocardial infarction/acute coronary syndrome, ischemic stroke, TIA, ventricular arrhythmia, or death from any cause
Time Frame: 90-days from presentation
Population: The data presented represents the total sample for intervention sites and control sites during the active implementation period.
Measure: Count of Participants; unit: Participants
Arm/Group | QI With External Facilitation | Control
Number analyzed (Participants) | 189 | 968
Participants | 16 | 96

3. Secondary Outcome: The Group Organization (GO) Score
Description: The GO Score refers to the Group Organization Score for improving TIA care quality; it is a measure of team activation and cohesion. The GO score is measured on a scale of 0-10 based on specific practices in place during a given time period and scored by the evaluation team. A score of 0-3 indicates the absence of a facility-wide approach; 4-5 reflects a developing facility-wide approach; 6-7 denotes basic proficiency with the presence of a comprehensive facility-wide program; and 8-10 indicates the presence of a mature, facility-wide system that can sustain key personnel turnover. The GO Score was measured only among the N=6 PREVENT sites.
Time Frame: Measured at the end of the one-year active implementation period
Population: The GO score is assessed at the facility level.
Measure: Mean (Standard Deviation); unit: units on the GO Score
Units Other Than Participants: Number of units (VA hospitals)
Groups:
- Active Implementation Sites: The six sites that actively implemented PREVENT.
Arm/Group | Active Implementation Sites
Number analyzed (Participants) | NA
Number analyzed (Number of units (VA hospitals)) | 6
units on the GO Score | 6.67 (1.374)

4. Secondary Outcome: Number of Quality Improvement Activities Completed
Description: The number of implementation activities completed during the one-year active implementation period
Time Frame: One-year active implementation period
Population: The six sites that implemented the PREVENT program
Measure: Mean (Standard Deviation); unit: number of activities per year
Units Other Than Participants: Number of units (VA hospitals)
Arm/Group | Active Implementation Sites
Number analyzed (Participants) | NA
Number analyzed (Number of units (VA hospitals)) | 6
number of activities per year | 26.5 (8.078)

5. Secondary Outcome: Program Satisfaction
Description: Overall staff satisfaction with the program was assessed with a single question with the response scale ranging from 1 to 7 where 7 indicated "extremely satisfied." Program satisfaction was measured only at the six PREVENT intervention sites.
Time Frame: Measured at the end of the one-year active implementation period
Population: Six PREVENT intervention sites
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of units (VA hospitals)
Arm/Group | Active Implementation Sites
Number analyzed (Participants) | NA
Number analyzed (Number of units (VA hospitals)) | 6
units on a scale | 6.23 (0.75)

ADVERSE EVENTS:
Time Frame: The active study period for each site was of variable duration ranging from 19-37 months; it began with the baseline interview and ended on September 2020.
Description: Adverse Events were monitored on a hospital level. Facility staff were the subjects of this research, the primary risk was breach of confidentiality which was not observed during the study period.
Arm/Group | QI With External Facilitation | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/36
Other Adverse Events (participants affected / at risk) | 0/6 | 0/36

LIMITATIONS AND CAVEATS:
PREVENT was implemented within VA facilities, which may limit generalizability. There may be diagnostic uncertainty when making a diagnosis of TIA. Because the intervention included multiple components, we are unable to estimate the unique associations of each specific element. Neither site selection nor allocation to waves was randomized. Although a 6-site sample provided adequate power for the detection of changes in processes of care, the study was not powered to detect changes in outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT02769338/Prot_SAP_000.pdf